CLINICAL TRIAL: NCT01828983
Title: Telephone Support During Overseas Deployment for Military Spouses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memphis VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda O. Nichols, Ph.D., Healthcare education specialist/Health Services Researcher, Memphis VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-11-2-0087
Record Dates: First submitted 2013-04-04; First posted 2013-04-11 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Military Personnel; Family Members; Resilience, Psychological; Deployment
Keywords: Telephone; Support groups; Social support; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone support groups (Experimental): Telephone support groups, each with participants and a trained group leader. Each hour-long telephone group will meet bi-monthly for six months for a total of 12 meetings. Groups are structured with education, skills building, and support. Participants will receive and use a Spouse Workbook with information and activities.
  Interventions: Behavioral: Telephone support groups
- Education webinars (Active Comparator): Education Webinar session topics are the same that are covered in the intervention arm without telephone interaction/support and skills building components. Each session is 30-minutes. Each participant receives a Spouse Workbook with information and activities.
  Interventions: Other: Education webinars

INTERVENTIONS:
Behavioral: Telephone support groups
  Arms: Telephone support groups
Other: Education webinars
  Arms: Education webinars

SUMMARY:
Deployment impacts both service member and family, and the cost can be high. Spouses' reactions to deployment may include emotional distress, loneliness, anticipatory fear or grief, somatic complaints, and depression. The goal is to help spouses learn ways to manage stress and solve problems related to deployment and reintegration, communication, managing long distance relationships, and other common problems. The study will compare telephone support groups to online education sessions. The study will enroll 160 spouses. In the Telephone Support groups, a group leader and participants will meet 12 times over six months to focus on education, skills building and support. Education Only online sessions will provide the same education content, without skills building or support. Content includes strategies to reduce or eliminate communication difficulties during deployment, how to find help; practical concerns during deployment; fostering resilience and decreasing stress; fostering relationships while apart, negotiating roles and relationships; changes during deployment; strategies to support the spouse and the service member; and cues to alert spouses when to seek mental health services for the family or themselves. Outcomes will include resilience, depression, anxiety and coping behaviors. Telephone data collection will be conducted at baseline, six and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* spouse or significant other (living as married for at least one year before deployment) of an overseas deployed military service member
* deployed at least six months

Exclusion Criteria:

* living as married for at least one year before deployment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda O Nichols, PhD, Principal Investigator — Memphis VA Medical Center and University of Tennessee Health Science Center; Jennifer L Martindale-Adams, EdD, Principal Investigator — University of Tennessee Health Science Center and Memphis VA Medical Center
Locations (1):
- Memphis VA Medical Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telephone Support Groups | Education Webinars
Started | 80 | 81
Completed | 80 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Support Groups | Education Webinars | Total
Number analyzed (Participants) | 80 | 81 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (8.4) | 35.5 (8.4) | 35.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 79 | 157
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 65 | 71 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 63 | 65 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 81 | 161

OUTCOME MEASURES:

1. Primary Outcome: Spouse Self-report of Resilience
Description: Connor-Davidson Resilience Scale (CD-RISC) measured at baseline, 6 and 12 months. Scores range from 0-100. Higher scores equal greater resilience.
Time Frame: Baseline, 6 months
Population: Participants who had data at baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Telephone Support Groups | Education Webinars
Number analyzed (Participants) | 80 | 81
units on a scale
  Resilience scores at baseline | 75.4 (1.3) | 75.9 (1.3)
  Resilience scores at 6 months: number analyzed (Participants) | 72 | 65
  Resilience scores at 6 months | 78.5 (1.1) | 81.0 (1.1)

2. Primary Outcome: Spouse Self Report of Anxiety
Description: Generalized Anxiety Disorder (GAD-7) measured at baseline, 6 and 12 months. Scores range from 0 to 21; higher scores equal more anxiety.
Time Frame: baseline, and 6 months
Population: Participants who had data at baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Telephone Support Groups | Education Webinars
Number analyzed (Participants) | 80 | 81
units on a scale
  Participants 'Anxiety baseline baseline scores | 6.0 (0.5) | 7.3 (0.5)
  Participants' Anxiety scores at 6 months: number analyzed (Participants) | 72 | 65
  Participants' Anxiety scores at 6 months | 5.3 (0.6) | 4.9 (0.6)

3. Primary Outcome: Spouse Self Report of Depression
Description: Patient Health Questionnaire - Depression (PHQ)-9 measured at baseline, 6 and 12 months. Scores range from 0-27 with higher scores indicating more depressive symptoms.
Time Frame: Baseline, 6 months
Population: Participants with data at baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Telephone Support Groups | Education Webinars
Number analyzed (Participants) | 80 | 81
units on a scale
  Participants' baseline scores | 5.5 (0.6) | 6.6 (0.6)
  Participants' scores at 6 months: number analyzed (Participants) | 72 | 81
  Participants' scores at 6 months | 3.8 (0.5) | 3.8 (0.5)

ADVERSE EVENTS:
Arm/Group | Telephone Support Groups | Education Webinars
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/81
Other Adverse Events (participants affected / at risk) | 0/80 | 0/81

LIMITATIONS AND CAVEATS:
There was no control arm where participants received no services. Participants were at various stages of the deployment process.

Lack of participation in the intervention was a study limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No